CLINICAL TRIAL: NCT03396172
Title: FreeDom : Innovative Strategy for the Management of COPD Exacerbations Combining Early Hospitalisation Discharge, Automated Oxygen Weaning at Home, Telemedicine and Tele-rehabilitation
Brief Title: FreeDom: Innovative Strategy for the Management of COPD Exacerbations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, François Lellouche, Principal Investigator, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21419
Record Dates: First submitted 2017-12-18; First posted 2018-01-10 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Oxygen Deficiency; COPD Exacerbation
Keywords: COPD; Homecare; Oxygen; Telemedicine; Automated oxygen adjustment; Rehabilitation program
MeSH Terms: conditions — Hypoxia; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): The intervention is an hospitalization with usual care. The hospitalization will take place in the usual setting and the hospital discharge will be decided by pulmonologists according to the usual criteria
  Interventions: Other: Control
- FreeDom (Active Comparator): FreeDom strategy (early discharge, automated weaning at home, telemedicine, telereadaptation):
  -initial conventional hospitalization before discharge home, O2 flow rate automatically titrated by FreeO2 (based on a SpO2 target). The hospital discharge will be possible if the definite criteria are met.
  After hospital discharge, patient will have home hospitalisation. Automated oxygen flow titration, patient education will be conducted for using the telemedicine system, for questionnaires and for the tele-rehabilitation program will be initiated for home hospitalization,
  Interventions: Device: FreeDom

INTERVENTIONS:
Other: Control — The hospitalization will take place in the usual setting and the hospital discharge will be decided by pulmonologists according to the usual criteria
  Other Names: Usual oxygen administration and usual hospitalization
  Arms: Control
Device: FreeDom — Early return home, patients using an innovative device that automatically adjusts and wean the oxygen flow (FreeO2 system) coupled to telemedicine and tele-rehabilitation
  Other Names: Early Hospital discharge with home hospitalisation
  Arms: FreeDom

SUMMARY:
The main objective of the study is to assess the "FreeDom" innovative strategy (FreeO2 at Domicile) to reduce hospitalization duration in patients with COPD exacerbation. This strategy associates early hospital discharge, automated O2 flow weaning with FreeO2 system, telemedicine and tele-rehabilitation.

The main hypothesis of this study is that the FreeDom strategy will reduce the number of hospitalization day by 50 percent at day 30.

DETAILED DESCRIPTION:
The main objective of the study is to assess the "FreeDom" innovative strategy (FreeO2 at Domicile) to reduce hospitalization duration in patients with COPD exacerbation. This strategy will enable an early return home, patients using an innovative device that automatically adjusts and wean the oxygen flow (FreeO2 system) coupled to telemedicine and tele-rehabilitation.

The main hypothesis of this study is that a strategy for an early return home with a home hospitalization managed by telemedicine will reduce the length of hospitalization by 50 percent from 30 days.

ELIGIBILITY:
Inclusion Criteria:

All patients hospitalized for COPD exacerbation for less than 48 hours will be considered.

* known or suspected COPD to entry
* Age > or = 40 years
* Ex-smoker history (10 pack / year or more)
* Acute Exacerbation: dyspnea of recent onset (less than 15 days)
* The need for oxygen therapy with a moderate rate: <6L / min to maintain SpO2 > 90% (for oxygen dependent patient, the oxygen flow must be higher than flow at home)

Exclusion Criteria:

* Refusal to consent to participate in the study,
* Indication for an imminent intubation according to the pulmonologist,
* Sleep Apnea
* NIV used at home
* Lack of FreeO2 system available at the time of randomization
* Non-autonomous and alone at home
* Patient alone at home
* Patients who live more than 50 km from the hospital
* Patient already included in the study within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-05-24 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The number of hospital days during COPD exacerbation at day 30. | 30 days
  The objective of the study is to reduced the hospitalisation days by 50 % at day 30 during COPD exacerbation

SECONDARY OUTCOMES:
Rate of Emergency consultation and hospital readmission | 1 and 3 months
  Rate of Emergency consultation and hospital readmission
Health Related Quality of Life | 1 and 3 months
  Survey of health related quality of life
Cost of care at 3 months | 3 months
  Economic evaluation about these 2 different strategy of COPD exacerbation management using micro-costing approach and including the cost of the FreeO2 technology
Oxygenation data (% of time in the SpO2 target, % of time with hypoxemia, % of time with hyperoxia) | From inclusion to hospital discharge and from hospital discharge to the end of oxygen therapy (around one week after discharge)
  The continuous measurement of SpO2 and O2 flow rate with the FreeO2 device (only in the FreeDom strategy) will allow the calculation of the % of time within the SpO2 target (recorded in the FreeO2) ± 2%, with hypoxemia (% of time with SpO2 < 85%) and with hyperoxia (% of time above SpO2 target +5%)
Number of consultations | 3 months
  Number of consultation : phone call, video consultation, rehabilitation, home visit

CONTACTS AND LOCATIONS:
Overall Officials: François Lellouche, Principal Investigator — Laval University
Locations (1):
- Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Canada